CLINICAL TRIAL: NCT03019354
Title: The Effect of Using High-flow Nasal Oxygen-delivery System in Patients Under Intravenous General Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201611036RIN
Record Dates: First submitted 2017-01-10; First posted 2017-01-12 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-04

CONDITIONS: Pulmonary Atelectases; Lung Injury; General Anesthesia
Keywords: high flow oxygen; pulmonary atelectasis; intravenous general anesthesia
MeSH Terms: conditions — Pulmonary Atelectasis; Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- high-flow nasal oxygen (Experimental): high-flow nasal oxygen was used during intravenous general anesthesia
  Interventions: Device: high-flow nasal oxygen
- Oxygen mask (Active Comparator): oxygen mask was used during intravenous general anesthesia
  Interventions: Device: Oxygen mask

INTERVENTIONS:
Device: high-flow nasal oxygen — Using high-flow nasal oxygen 10 L/min before anesthesia induction, then using high-flow nasal oxygen 30-50 L/min during intravenous general anesthesia.
  Other Names: High-flow nasal cannula
  Arms: high-flow nasal oxygen
Device: Oxygen mask — Using oxygen mask with oxygen flow 10 L/min before and during intravenous general anesthesia.
  Arms: Oxygen mask

SUMMARY:
In general anesthesia, gas exchange was altered by shunt and uneven ventilation perfusion ratios. Lung atelectasis was a cause of impaired oxygenation. High-flow nasal cannula oxygen therapy delivers adequately heated and humidified medical gas at up to 60 L/min of flow. It has physiological effects: reduction of anatomical dead space, positive end expiratory pressure (PEEP) effect, constant fraction of inspired oxygen, and good humidification. The hypothesis of this study is using high-flow nasal oxygen in intravenous general anesthesia could improve lung function and prevent lung atelectasis.

DETAILED DESCRIPTION:
After general anesthesia, almost 90% patients have lung atelectasis. The lung atelectasis persisted even after the surgery, and caused post operative complication, for example: fever, pleural effusion, hypoxemia, pneumonia, and respiratory failure. So, how to improve lung function after the surgery is a important issue. High-flow nasal cannula oxygen therapy delivers adequately heated and humidified medical gas at up to 60 L/min of flow. It provides respiratory support: 1. Reduction of dead Space by clearance of expired air in the upper airways. 2. Delivering positive airway pressure. 3. delivering optimal humidity, which helps maintain function of the mucociliary transport system, clearing secretions and reducing the risk of infections. Many reports suggest that high-flow nasal cannula decreases breathing frequency and work of breathing and reduces intubation rate in critical ill patients. Although high-flow nasal cannula was used widely in intensive care unit (ICU) , there are no enough evidence in patients under general anesthesia. The hypothesis of this study is that using high-flow nasal oxygen in intravenous general anesthesia could improve lung function and prevent lung atelectasis. Liver tumor radiofrequency ablation was performed sometimes in patients under general anesthesia. Intravenous general anesthesia is one of the anesthesia choice. Oxygen mask is the traditional oxygen delivery system. Apnea, hypoxemia, and CO2 retention are common situation in intravenous general anesthesia. So high-flow nasal oxygen is an ideal oxygen delivery system in intravenous general anesthesia. This randomized control study will enroll patients receiving CT guided liver tumor radiofrequency ablation under general anesthesia. One group will receive high-flow nasal oxygen, the other group will receive traditional oxygen mask. The primary outcome is lung atelectasis area in CT scan. The secondary outcome is respiratory function (for example: arterial blood gas, lung injury biomarkers, saturation, postoperative pulmonary complication)

ELIGIBILITY:
Inclusion Criteria:

* Patients with hepatic tumor undergoing CT guided radiofrequency ablation
* Age > 20 years old

Exclusion Criteria:

* Cardiac dysfunction, such as heart failure > NYHA class II, coronary arterial disease
* Impaired renal function, cGFR< 60 ml/min/1.73 m2
* Pulmonary disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Chest CT image atelectatic area | At the end of surgery
  lung atelectasis (-100 to +100 Hounsfield Unit) was calculated and as percent of the total area of the lung at the basal scan.

SECONDARY OUTCOMES:
postoperative pulmonary complications | within the first 7 days after surgery
  postoperative pulmonary complications including pneumonia, pleural effusion, and acute lung injury.
lung injury | At the end of surgery
  lung injury biomarkers including Clara cell protein, Plasma neutrophil elastase.

OTHER OUTCOMES:
Respiratory gas exchange function | At the end of surgery
  blood gas analysis including PaO2, PaCO2
need for supplemental oxygen therapy | within the first 7 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Yu Wu, MD,PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shih CC, Liang PC, Chuang YH, Huang YJ, Lin PJ, Wu CY. Effects of high-flow nasal oxygen during prolonged deep sedation on postprocedural atelectasis: A randomised controlled trial. Eur J Anaesthesiol. 2020 Nov;37(11):1025-1031. doi: 10.1097/EJA.0000000000001324. PMID 32890016